CLINICAL TRIAL: NCT05517460
Title: The Efficacy of Auricular Acupressure on Improving Constipation Among Residents in Community Rehabilitation Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Huang, Hui-Chuan, The Efficacy of Auricular Acupressure on Improving Constipation among Residents in Community Rehabilitation Center, Taipei Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 202204021
Record Dates: First submitted 2022-08-19; First posted 2022-08-26 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia; Constipation
MeSH Terms: conditions — Schizophrenia; Constipation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group I(auricular acupressure and usual care) (Experimental): Experimental group I receives 8 weeks of auricular acupressure first, then interventions are stopped for two month as residual effect wash-out period. And after that Experimental group I receives 8 weeks of routine health care of constipation.
  Interventions: Other: Auricular acupressure; Other: health education
- experimental group II(usual care and auricular acupressure) (Experimental): Experimental group II receives 8 weeks of routine health care of constipation first, then interventions are stopped for two month as residual effect wash-out period. And after that Experimental group II receives 8 weeks of auricular acupressure .
  Interventions: Other: Auricular acupressure; Other: health education

INTERVENTIONS:
Other: Auricular acupressure — The participant in Intervention period will receive acupressure on ear Shenmen point, ear Large intestine point, ear Rectumn point and ear San Jiao point.
Other: health education — health education for self-care and medication adherence

SUMMARY:
The purpose of the study is to examine the effect of auricular acupressure on improvement of constipation and heart rate variability among residents with schizophrenia in community rehabilitation Center.The hypothesis of this study is that residents with schizophrenia in Community Rehabilitation Center receiving auricular acupressure can improve the symptoms of constipation and heart rate variability.By identifying the effectiveness of auricular acupressure can reduce the occurrence of constipation; suitable care can be suggested to improve gastrointestinal health in residents of Schizophrenia in community rehabilitation center.

DETAILED DESCRIPTION:
Due to the use of psychiatric medication and the impairment of cognition lead to poor lifestyle which is result in constipation among the residents of community rehabilitation center.In addition, the residents affected by psychosis and poor cognition are hard to pay attention and implement on the non-pharmacological interventions completely with complicated process.Therefore, contriving a simple intervention, which may improve constipation and constipation-related symptoms. The purpose of this study is to examine the effectiveness of applying auricular acupressure for relieving the constipation symptoms of residents of Schizophrenia in community rehabilitation center. A cross-over study design is used for this study. The eligible participants were random assign to experimental group I or experimental group II. Experimental group I received 8 weeks of auricular acupressure then 8 weeks of routine health care of constipation. Experimental group II received same interventions in reverse order (8 weeks of routine health care of constipation then 8 weeks of auricular acupressure).In both groups, any interventions were stopped for two month as residual effect wash-out period after 8 weeks intervention. Outcome measures include demographic variables, general health status and defecation condition. Subjective defecation condition is related to self-perceived constipation measured by the Patient Assessment of Constipation Symptoms scale. Objective defecation condition includes frequency of defecation, the grade of Bristol Stool Scale and heart rate variability. Mean, standard deviation, frequency, percentage, t-test and chi-square test will be used to analyze the data. In addition, generalized estimating equations will be used to examine the effect of auricular acupressure on improving constipation. By identifying the effectiveness of auricular acupressure can reduce the occurrence of constipation; suitable care can be suggested to improve gastrointestinal health in residents of Schizophrenia in community rehabilitation center.

ELIGIBILITY:
Inclusion Criteria:

* Living in community rehabilitation center for at least six months and above.
* Community rehabilitation center residents aged 40 and over.
* Clinical diagnosis of Schizophrenia.
* Having constipation-related symptoms: meet at least one of the following conditions:

  1. Chief complaint of discomfort of defecation such as difficulty in defecation, hard stool, straining during defecation, feeling of incomplete defecation, feeling of obstructed defecation, defecation frequency less than three times a week.
  2. Objective symptoms: Type 1 or 2 of Bristol Stool Form assessment.
  3. Long-term use(1 month and above) of laxatives such as MgO、Sennoside etc ., or need to use an enema to defecate.

Exclusion Criteria:

* Incapable of complying with the direction and responding to questionnaires.
* Having wound or local skin lesion on acupressure point.
* Having organic constipation caused by abdominal operation in the past.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Patient Assessment of Constipation Symptoms questionnaire | Baseline
  Patient Assessment of Constipation Symptoms
Patient Assessment of Constipation Symptoms questionnaire | at eight weeks after intervention
  Patient Assessment of Constipation Symptoms
Bristol Stool Scale | Baseline
  frequency of defecation, range of 1-7 and low score indicate constipation
Bristol Stool Scale | at four weeks after intervention
  frequency of defecation, range of 1-7 and low score indicate constipation
Bristol Stool Scale | at eight weeks after intervention
  frequency of defecation, range of 1-7 and low score indicate constipation
heart rate variability. | Baseline
  heart rate variability.
heart rate variability. | at four weeks after intervention
  heart rate variability.
heart rate variability. | at eight weeks after intervention
  heart rate variability.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chuan Huang, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei County, Taiwan